CLINICAL TRIAL: NCT06231641
Title: The Effects of Lemborexant on the Ability to Sleep During Daytime: A Feasibility Study to Evaluate the Potential of Lemborexant to Treat Shift Work Disorder
Brief Title: The Effects of Lemborexant on the Ability to Sleep During Daytime
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Alex Desautels, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DVG-IIS-M001-1008
Record Dates: First submitted 2024-01-17; First posted 2024-01-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Shift-Work Sleep Disorder
Keywords: Daytime sleep episodes; Polysomnographic recordings; Subjective sleep evaluations; Total sleep time (TST); Wake after sleep onset (WASO)
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — lemborexant

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled crossover mono-centric feasibility study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active treatment condition (Active Comparator): Lemborexant at a 5mg dose is delivered in a film-coated tablet
  Interventions: Drug: Lemborexant 5 MG [Dayvigo]
- Placebo condition (Placebo Comparator): Placebo is delivered in a film-coated tablet
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Drug: Lemborexant 5 MG [Dayvigo] — Lemborexant 5 mg will be taken orally once per day just prior to initiating laboratory-supervised daytime sleep episodes, for three consecutive days, within a few minutes before going to bed, with at least seven hours remaining before the planned time of awakening.
  Arms: Active treatment condition
Other: Matching Placebo — Matching placebo will be taken orally once per day just prior to initiating laboratory-supervised daytime sleep episodes, for three consecutive days, within a few minutes before going to bed, with at least seven hours remaining before the planned time of awakening.
  Arms: Placebo condition

SUMMARY:
This study aim to evaluate whether a dose of 5 mg of lemborexant, as compared to a placebo, may improve daytime recovery sleep, without producing lingering sleepiness during wakefulness, using a 3-day simulated night shift protocol in the lab under constant monitoring.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed conset will undergo 2 screening visits to determine eligibility for study entry. Selected participants will then stay twice in the lab (active treatment condition and placebo condition), each visit lasting approximately 4 days. Participants will stay awake across the night and sleep during the day. Only the experimental condition will be different between the two visits (lemborexant or placebo). These experimental visits will be double-blind, in counterbalanced order and separated by an interval of at least 2 weeks (washout period).

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill all of the following inclusion criteria to be eligible for inclusion in this study:

1. Men or women aged between 20 and 65 years, inclusive
2. Be willing and able to give informed consent for study participation
3. Participants must not have done shiftwork in the past year
4. Normal vital signs values are: oral body temperature between 36.1 and 37.5 ºC (95 and 99.5 °F), supine SBP between 90 and 140 mmHg inclusive; supine DBP between 55 and 90 mmHg inclusive; heart rate between 50 and 100 bpm inclusive.
5. Be willing to comply with all study requirements and procedures for the duration of the study, including refraining from consuming alcohol 48 hours prior to each experimental visit and grapefruit products (juice or fruit itself), Seville orange, lime, pomelo, carambola and pomegranate during all the duration of the study (from Visit 1 to Visit 4).
6. Women who:

   * Are postmenopausal, with amenorrhea for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If of childbearing potential agree to practice effective double barrier methods of contraception, from the time of the signing of informed consent through the last dose of study drug and for 30 days after dosing stops (1 ovulatory cycle), or agree to completely abstain from intercourse.

   Men with women partners of childbearing potential are also expected to practice effective barrier methods of contraception from the time of signing informed consent through the last dose of study drug and for 30 days after dosing stops.
7. Self-reported bedtime was between 9 pm and midnight on 4-7 nights per week.

Exclusion Criteria:

Participants must not meet any of the following exclusion criteria:

1. Body mass index > 32 as calculated from the participant's height (m) and weight (kg); weight (kg)/square height (m²)
2. Presence of a sleep disorder, such as a diagnosis of insomnia, narcolepsy, sleep paralysis, active somnambulism (history of childhood somnambulism is accepted), hypnagogic/ hypnopompic hallucinations, and REM behavior disorder, will be excluded based on the clinical interview. For sleep apnea syndrome, an apnea-hypopnea index > 15 per hour of sleep on the first screening night will be used as an exclusion criterion. For periodic limb movement disorder, an index of periodic limb movements during sleep associated with an arousal > 15 per hour of sleep on the first screening night will be used as an exclusion criterion.
3. History of epilepsy
4. Any previous serious head injury or stroke
5. Any evidence of psychiatric disorder (including Beck Depression Inventory [BDI] ≥ 20 at screening, or a score of 3 on item related to suicidal ideas)
6. Evidence of any clinically significant, or unstable, acute or chronically progressive medical or surgical disorder (including planned medical procedures that may impact sleep), or any condition that may interfere with the absorption, metabolism, distribution, or excretion of the study drug, or may affect the participant's safety
7. Clinically significant and abnormal electrocardiogram (ECG; including QTc ≥ 450 ms for males, 460 ms for females) or a history of cardiovascular disease including poorly controlled hypertension, ischemic heart disease, arrhythmia, or severe heart failure
8. Severe hepatic impairment
9. Positive qualitative urine drug screen (opiates, cocaine, amphetamine, cannabinoids, barbiturates, phencyclidine, benzodiazepines, methadone, propoxyphene) and alcohol test (breathalyzer), at screening and before each experimental visit
10. Current use of medications that are moderate or strong CYP3A4 inhibitors or inducers or CYP2B6 substrates (Appendix 1)
11. Use of any substance with psychotropic effects or properties known to affect sleep/wake, including hypnotics, neuroleptics, opioid derivatives, antihistamines, stimulants, antidepressants, within one week or five half-lives (whichever is longer) prior to PSG screening
12. Use of any over-the-counter sleep medications including tryptophan, valerian root (Valeriana officinalis), kava (Piper methysticum Forst), melatonin, St John's Wort (Hypericum perforatum), Alluna (herbal sleep supplement with valerian root), and hemp within one week or five half-lives (whichever is longer) prior to screening
13. Consumption of xanthine-containing beverages (i.e., tea, coffee, or cola) of more than 5 cups or glasses per day
14. Participation in any other trial within 30 days before the screening visit
15. Any travel across more than one time zone in the month prior to screening at any time during the study
16. Other exclusion criteria based on adverse events (AE) or serious adverse events (SAE) reported in the Investigator Brochure
17. Women who are pregnant, during the study or within one month after the study, or are breastfeeding
18. Individuals may be excluded from participating in the study based on the clinician's judgement.
19. Participants with lactose or galactose intolerance (galactosemia or glucose-galactose malabsorption)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Total sleep duration (objective measure) | during the intervention
  Assess the efficacy of lemborexant compared to placebo on PSG measured total sleep time (TST) during daytime recovery sleep using the mean data of the second and third daytime sleep episodes in each condition.
Wake after sleep onset (objective measure) | during the intervention
  Assess the efficacy of lemborexant compared to placebo on polysomnographically (PSG) measured wake after sleep onset (WASO) during daytime recovery sleep using the mean data of the second and third daytime sleep episodes in each condition

SECONDARY OUTCOMES:
Total sleep duration (subjective measure) | during the intervention
  Evaluate the participant-reported daytime recovery sleep quality, measured as subjective TST (sTST), under lemborexant in comparison to placebo using the mean data of the second and third daytime sleep episodes in each condition
Wake after sleep onset (subjective measure) | during the intervention
  Evaluate the participant-reported daytime recovery sleep quality, measured as subjective WASO (sWASO), under lemborexant in comparison to placebo using the mean data of the second and third daytime sleep episodes in each condition.

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS du Nord de l'ile de Montreal (CIUSSS-NIM) - Hôpital du Sacré-Cœur de Montréal (HSCM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No